CLINICAL TRIAL: NCT04328142
Title: Effectiveness of Qigong vs. Physiotherapy to Improve Quality of Life of Women With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Effectiveness of Qigong vs. Physiotherapy to Improve Quality of Life of Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Abel Mejías Gil, PHYSIOTHERAPIST, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11//2012
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Physiotherapy; Qigong; Quality of life
MeSH Terms: conditions — Fibromyalgia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Participants were randomized to a Qigong exercise programme group, a Physiotherapy treatment group and control group for a 6 week study.
Who Masked: Outcomes Assessor
Masking Description: Neither the participants nor their therapists were blind to the treatment allocation. However, the assessor was independent to the study and was not aware of the treatments applied or the objective of the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qigong (Experimental): The Qigong experimental group performed the 20 figures to improve health and longevity described by the master of Qigong 'Wang Ziping'. These are based on therapeutic exercises of Traditional Chinese Medicine. They work on breathing, flexibility and balance. Each figure was repeated 6 times. The sessions were administered twice a week during 45 minutes and were guided by a Doctor in Western Medicine who is also qualified as a Doctor of Traditional Chinese Medicine and Qigong teacher.
  Interventions: Other: Qigong group
- Physiotherapy (Experimental): The physiotherapy experimental group completed an active exercises program guided by a qualified physiotherapist. The exercise programme was based on active shoulder, hips and spine kinesiotherapy. It included a warm up of 3-5 minutes walking, followed by 6 repetitions of shoulder and hip exercises in standing, cervical spine exercises in sitting or standing, according to the comfort of the patient, thoracic and lumbar spine exercises performed in supine on a mat and balance exercises in standing. Stretching exercises were also performed at the end of the session. The exercises were accompanied by gentle breathing coordinated with the movements. The sessions were administered twice a week during 45 minutes.
  Interventions: Other: Physiotherapy
- Control (No Intervention): The control group did not receive any intervention. The participants continued with their routine medical treatment.

INTERVENTIONS:
Other: Qigong group — Traditional Chinese Medicine exercise programme
  Arms: Qigong
Other: Physiotherapy — Physiotherapy exercise programme
  Arms: Physiotherapy

SUMMARY:
This study analyze the effectiveness of a Physiotherapy treatment versus a Qigong exercise programme improving quality of life of subjects with Fibromyalgia.

DETAILED DESCRIPTION:
Objective:

This study investigated the effectiveness of a Physiotherapy treatment versus a Qigong exercise programme for the improvement of the quality of life of subjects with Fibromyalgia.

Design:

A single-blind randomized clinical controlled trial.

Setting:

University of Extremadura, Spain

Subjects:

Women with Fibromyalgia

Interventions:

141 Participants were randomized to a Qigong exercise program group (n=47), a physiotherapy treatment group (n=47) and control group (n=47) for 6 weeks.

Main Measures:

Measures were taken at baseline (week 0), pre intervention (week 1) and post intervention (week 6). The primary outcome measure were quality of life (Spanish Fibromyalgia Impact Questionnaire (SFIQ), pain (VAS), perceive exertion (Borg scale), spirometry measures (Spirobank-G MIR spirometry) and balance (Wii-Fit, Nintendo ©). The secondary outcome measures were flexibility (Wells and Dillon test and Sit and Reach test), Range of movement (goniometer), muscle strength (Lowett scale).

ELIGIBILITY:
Inclusion Criteria:

* women between 30 and 65 years old,
* diagnosed with Fibromyalgia by a specialized physician,

Exclusion Criteria:

* The exclusion criteria were to present any limitation of mobility due to Fibromyalgia or other pathology, previous practice or knowledge of Qi gong, to be under Physiotherapy treatment and to practice any physical exercise.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

PRIMARY OUTCOMES:
Change from the Spanish Fibromyalgia Impact Questionnaire (SFIQ) at post intervention (week 6) | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  SFIQ measures the level of quality of life of subjects with Fibromyalgia with a score of 0 to 100. A higher score indicates more impact of the condition on the life of the person and therefore less quality of life.
Change from Visual Analogue Scale (VAS) at post intervention (week 6) | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  The Visual analogue scale measures the level of pain with a score of 0 to 10 where 0 indicates no pain and 10 indicates maximun pain.
Change from Borg Scale of perceived exertion at post intervention (week 6) | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Borg scale measures the perceived exertion of a subject with a score of 0 to 10 where 0 is the minimum exertion and 10 is the maximun exertion.
Changes from the values registered by the Spirobank-G (MIR)® spirometer | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Spirometry measures respiratory values being the reference values (Knudson model) for a 50 year old woman with 1,65 cm of height and 65 kilos weight: FVC (Forced vital capacity)= 3.611, FEV1 (Forced expiratory volume) = 2.7505, FEV1%= 76.17%, FEF (Forced expiratory flow) 25-75%= 2.625, PEF (peak expiratory flow)= 6.222
Change from the centre of gravity registered with Wii-fit Nintendo® | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Static balance and postural control is the ability to maintain the centre of gravity within the base of support. Centre of gravity is measured in percentage through posturography study. A higher percentage means better balance
Change from the monopodal stance test registered with Wii-fit Nintendo® | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Monopodal stance test measures static balance in percentage through posturography study. It is measure in percentage from 0 to 100 and a higher percentage means a better result.

SECONDARY OUTCOMES:
Change from range of movement measured with goniometer | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Shoulder and hip range of movement
Change from muscle strength measured with Lovett scale | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Shoulder and hip range of movement.Lovett scale is a modification of Daniels and Worthingham. The scale is measured from 0 to 5 where 0 means no muscle activation strength and 5 means normal strength against resistance
Change from flexibility measured with the Wells y Dillon scale | Baseline (week 0), pre intervention (week 1) and post intervention (week 6).
  Flexibility is measured with this scale with the patient sitting and reaching the feet. It is measured in centimeter and a more positive value means a better record.

IPD SHARING:
Plan to Share IPD: No